CLINICAL TRIAL: NCT05033379
Title: Impact of Circadian Alignment, Autonomic Control, and Physiologic Feedback on Measures of Resilience: A Multicenter Randomized Controlled Trial
Brief Title: Healthcare Worker Resilience as Measured by Physiologic Feedback
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Cindy Kin, Assistant Professor of Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 61917
Record Dates: First submitted 2021-08-17; First posted 2021-09-02 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Burnout, Professional
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Experimental): Instruction about importance of sleep.
  Interventions: Behavioral: Control
- Coaching (Experimental): Undergo resilience coaching
  Interventions: Behavioral: Resilience coaching

INTERVENTIONS:
Behavioral: Control — Importance of sleep
  Arms: Control Arm
Behavioral: Resilience coaching — Arena Strive
  Arms: Coaching

SUMMARY:
Reliably achieving peak performance requires balancing the strain of the prior day with sufficient recovery to be ready for the next day. Surgery has a long standing tradition long hours of hard work often at the expense of adequate sleep. Decreased sleep and recovery has physiologic consequences which can be measured using biometric data. The goal of this study is to quantify surgeon performance and biometric data to understand how modifiable behaviors including mindfulness training and diet can maximize recovery and performance. The goal of this study is to quantify the impact if modifiable daily behaviors including sleep, nutrition, in order to understand the factors that contribute to high level performance, burnout, and physician wellbeing in surgical trainees and attendings.

DETAILED DESCRIPTION:
Informed consent will be obtained prior to participation in the research study. A member of the research team will provide the participant with the consent form and allow them adequate time to read and ask questions prior to giving consent. If consent is not obtained, the participant will not be allowed to participate in the research study.

Participants will be asked to wear a biometric sensor for six months. The biometric sensor (The WHOOP strap) collects heart rate, heart rate variability, activity, and sleep metrics. Half of the participants will complete coaching to improve resilience with Arena Strive and half will be a control group instructed that sleep is important. In the latter 3 months of the study, the control group will have the opportunity to wear a continuous glucose monitor. At the completion of the study period all participants will have access to Arena strive coaching.

Other data gathered will be in the form of surveys and comments from subjects on wellness, burnout, modifiable activities including sleep, nutrition, glucose levels using continuous glucose monitoring, exercise and mindfulness.

ELIGIBILITY:
Inclusion Criteria:

* Study participants will include full time clinically active healthcare workers

Exclusion Criteria:

* Exclusion criteria will be anyone who is not a full-time clinical healthcare worker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-08-29 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Recovery | 6 months
  Using WHOOP algorithm, recovery will be quantified using heart rate variability and sleep, and serve as a measure of stress and resilience

SECONDARY OUTCOMES:
Burnout | 6 months
  The Physician Fulfillment Index is a quantitative measure of physician burnout and will be administered at baseline and at the end of the study.
Health Habits | 6 months
  Changes in sleep metrics (duration of sleep, quality of sleep, and pre-sleep habits including light exposure and eating habits before sleep) and diet habits (evaluated by dietary pattern, ie, traditional Westernized, healthy Mediterranean, unhealthy - animal protein and alcohol, at beginning and end of the study) will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Health Care, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No